CLINICAL TRIAL: NCT01753778
Title: A Prospective Non-Randomized Unblinded Study Evaluating Treatment of Forefoot Pain Related to Nerve Entrapment Using the Cryo-Touch III Device
Brief Title: Study Evaluating Treatment of Forefoot Pain Related to Nerve Entrapment Using the Cryo-Touch III Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MYO-0614
Record Dates: First submitted 2012-12-14; First posted 2012-12-20 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Entrapment Neuropathy
Keywords: Nerve Entrapment, Morton's neuroma, entrapment neuropathy
MeSH Terms: conditions — Charcot-Marie-Tooth Disease; Nerve Compression Syndromes; Morton Neuroma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Treatment with Cryo-Touch III Device at Day 0
  Interventions: Device: Cryo-Touch III Device

INTERVENTIONS:
Device: Cryo-Touch III Device — Treatment with Cryo-Touch III

SUMMARY:
A proof of concept study to evaluate the feasibility of safe and effective treatment through optimization of the Cryo-Touch III Device for temporary relief of pain.

DETAILED DESCRIPTION:
Over 100 million patients in the United States suffer from chronic pain. Chronic pain conditions are often debilitating, taking a toll on a patient's physical and mental welfare. Though a variety of pain management techniques currently exist, the most common nonsurgical options provide slow-acting and/or short-term relief. Medication, often in the form of non-steroidal anti-inflammatory drugs (NSAIDs) and opioids, comes with an array of side effects such as nausea and vomiting. Medication also presents the possibility of more serious effects such as increased risk of heart attack and stroke, and tolerance or dependency issues. Surgical strategies tend to be reserved for more severe cases and are limited by the risks and complications typically associated with surgery including bleeding, bruising, scarring, and infection. A nonsurgical, minimally invasive, long-lasting approach to chronic pain management is desirable.

Myoscience, Inc. (Redwood City, CA) has developed a pain management device - the Cryo-Touch III - for a novel, minimally invasive procedure using focused cold therapy to target sensory nerve tissue and offer long-lasting pain relief through cryoanalgesia. The device operates on the well-established cryobiology principle that localized exposure to controlled, moderately, low temperature conditions can alter tissue function. The therapy treats nerves via a probe in the form of an assembly of small diameter needles, creating a highly localized, low temperature treatment zone around the probe. This focused cold therapy creates a conduction block that prevents nerve signaling. Prior studies of the Cryo-Touch, Cryo-Touch II, Cryo-Touch III (a.k.a. PCP 1.0) devices have provided preliminary evidence of effectiveness on motor nerves and have been shown to be safe with no serious device-related adverse events.

Though studies have proven efficacious in targeting motor nerves, the device's effect on sensory nerves has yet to be investigated in the clinical setting. The goal of the study described herein is to evaluate the degree and duration of effect of the Cryo-Touch III in reducing chronic pain by targeting sensory nerves.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 years of age and older. Female subjects of childbearing potential must not be pregnant at time of treatment.
2. Trial participants must have a confirmed diagnosis of pain in the forefoot that is due to entrapment of related nerves.
3. Any medication must be maintained on a stable schedule for at least two weeks prior to treatment. No washout period is allowed.
4. Must have an average score for pain of ≥ 4/10 Visual Analog Scale (VAS) over the last 7 days.
5. Subject is willing and able to give written informed consent and able to comply with study instructions.
6. Subject is willing and able to comply with study instructions and commit to all follow-up visits for the duration of the study.
7. Subject is in otherwise good general health and free of any systemic disease state or physical condition that might impair evaluation or which in the investigator's opinion, exposes the subject to an unacceptable risk by study participation.

Exclusion Criteria:

1. History of fibromyalgia, cerebrovascular accident (CVA), foot or lower limb trauma, stroke, or bone deformity.
2. Patient who has severe pain for any reason other than forefoot pain due to nerve entrapment.
3. Any additional diagnosis that in the opinion of the investigator directly contributes to forefoot pain.
4. Any concomitant inflammatory disease or other condition that affects the joints (e.g. rheumatoid arthritis, metabolic bone disease, gout, active infection, etc.)
5. Surgical invention previously conducted in the forefoot area.
6. Any injection (neurolytic, sclerosing, anesthetic, etc.) to the foot within the last 2 months.
7. Any use of systemic injections (in any area) for pain management within the last 4 months.
8. Any use (i.e. oral, topical, inhaled and/or injected) of anesthetics or steroids within the last 30 days.
9. Current enrollment in an investigational drug or a device study that specifically targets pain treatment.
10. Enrollment in any other investigational drug or device study or participation within the last 30 days.
11. Any clotting disorder and/or use of any anticoagulant (e.g., warfarin, clopidogrel, etc.) within seven (7) days prior to administration of the treatment.
12. Allergy or intolerance to any preparatory treatment agent or any other substance utilized within the study.
13. Any local skin condition at the treatment site that in the investigator's opinion would adversely affect treatment, outcomes, or subject safety.
14. Any confounding diagnosis or medical condition that in the investigator's opinion would adversely affect study participation or subject safety.
15. Any chronic medication use (prescription, over-the-counter, supplements, etc.) that in the investigator's opinion would adversely affect study participation or subject safety.
16. Any reason that, in the opinion of the investigator, the subject may not be a suitable candidate for study participation (i.e., history of noncompliance, drug dependency, any related foot injury due to a worker's compensation claim, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-11; Primary Completion 2013-05 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Improvement of forefoot pain at day 7 | 7 days
  Improvement of forefoot pain due to nerve entrapment, as measured on the Visual Analog Scale (VAS) for pain at Day 7 as compared to baseline (Day 0).

SECONDARY OUTCOMES:
Duration of Treatment | 56 days
  Duration of Treatment Effect/No Effect
Safety Endpoints | 56 days
  Adverse events and SAEs/UADEs will be assessed at all visits. Incidence of serious adverse events (SAEs) and unanticipated adverse device effects (UADEs) will be recorded. A serious adverse event is one that meets the ISO definition of SAE

CONTACTS AND LOCATIONS:
Overall Officials: Srinivas Nalamachu, MD, Principal Investigator — International Clinical Research; Jonah Mullens, DPM, Principal Investigator — SOAR Medical Group
Locations (2):
- United States (2):
  - SOAR Medical Group, Redwood City, California
  - International Clinical Research, Overland Park, Kansas